CLINICAL TRIAL: NCT03719859
Title: Multicenter Randomized Trial of Home vs. Physical Therapist-Directed Rehabilitation for Reverse Total Shoulder Arthroplasty
Brief Title: Home Exercise vs PT for Reverse Total Shoulder Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Orthopedic Research and Education Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18082102
Record Dates: First submitted 2018-10-16; First posted 2018-10-25 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Shoulder Arthritis; Rotator Cuff Tear Arthropathy
Keywords: reverse total shoulder arthroplasty; physical therapy
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy | interventions — Physical Therapy Modalities; Home Infusion Therapy

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to one of two groups (surgeon directed home therapy or formal physical therapy). If subjects in either group are dissatisfied with the outcome of their rehabilitation process, they will be afforded the opportunity to cross-over to the other arm of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Therapy (PT) Group (Experimental): Subjects will attend formal physical therapy after surgery.
  Interventions: Other: Physical Therapy
- Home Therapy (HT) Group (Active Comparator): Subjects will receive instruction from clinical staff regarding home therapy exercises after surgery.
  Interventions: Other: Home Therapy

INTERVENTIONS:
Other: Physical Therapy — Subjects who will participate in the physical therapy intervention group will attend therapy 4-6 days after discharge from the hospital, and continue in therapy approximately once a week for three months. The physical therapy progression will follow the standard of care developed at Duke Sports Medicine Physical Therapy for rehabilitation following RSA. Some of the patients in the PT intervention cohort may have physical therapy at an institution outside of Midwest Orthopaedics at Rush. All patients, whether in the Rush system or outside, will be given a prescription with the identical instructions for "physical therapy, status post (R/L) reverse total shoulder arthroplasty, 1-2 x per week x 12 weeks."
  Other Names: PT
  Arms: Physical Therapy (PT) Group
Other: Home Therapy — The surgeon/Nurse Practitioner/Physician Assistant will advance rehabilitation exercises and activity guidelines at customary scheduled postoperative appointments for this surgical procedure: 2 weeks (+/- 5 days), 6 weeks (+/- 1 week), 3 months and 6 months (+/- 1 month), and 1 and 2 years (+/- 2 months).
  Other Names: HT
  Arms: Home Therapy (HT) Group

SUMMARY:
The primary objective of this study is to compare outcomes between formal clinic based physical therapy (PT) rehabilitation and surgeon directed home therapy (HT) after reverse total shoulder arthroplasty (RSA) as measured by pain, range of motion, Single Assessment Numerical Evaluation (SANE), and American Shoulder and Elbow Surgery (ASES) scores at 6 weeks, 3, 6, 12, and 24 months postoperatively. The secondary objective of this study is to determine if PT rehabilitation following RSA is associated with a higher level of postoperative complications, specifically acromial stress fractures or dislocation. This information will be useful to discern if PT is effective in providing pain relief more quickly, as well as improved motion and self-reported functional outcomes following RSA, which can assist surgeons and rehabilitation specialists in designing optimal care plans for this patient population. The project will also help to clarify if PT services place patients who have RSA at higher risk for acromial stress fractures or dislocation.

DETAILED DESCRIPTION:
Reverse total shoulder arthroplasty (RSA) is a relatively new solution for the patient with osteoarthritis of the glenohumeral joint with a deficient rotator cuff, or patients with glenohumeral osteoarthritis with excessive erosion of the posterior glenoid. Since the approval of RSA in 2003, the utility has increased such that this procedure represented 33% of all shoulder arthroplasties performed in the United States in 2011, and represents greater than 90% in some European countries The RSA prosthesis is effective at providing improved active motion and function due the semi-constrained design--substituting for the centering effect of the rotator cuff and allowing the deltoid to elevate or abduct the arm with fixed-fulcrum kinematics without a functional rotator cuff. Many factors influence the potential for successful outcome following RSA: proper patient selection, surgeon experience level, prosthesis characteristics, surgical technique and approach, and postoperative rehabilitation. Prior researchers have explored the effect of surgical technique, type of prosthesis, and surgery indications on outcome following RSA, however there is no data published on the impact of postoperative rehabilitation following this surgery.

A systematic review of the literature reveals that complications following RSA occur with four times greater incidence than complications following anatomic total shoulder arthroplasty (TSA). Complications following RSA which may be impacted by the exercises associated with physical therapy include instability and acromion stress fractures. A systematic review of the literature was conducted to determine if complication rates following RSA differ due to surgical approach, type of prosthesis (medialized or lateralized center of rotation), and the indication for the procedure. The authors of this review acknowledge that postoperative rehabilitation can impact the clinical and functional outcome of RSA and complication rate, however did not study this variable due to the heterogeneous approach to rehabilitation for the multi-center study.

Experts in the field of shoulder rehabilitation have published clinical guidelines for rehabilitation following reverse shoulder arthroplasty. One set of published guidelines is based on biomechanical and basic science healing timeframes associated with the tissue attrition following RSA. The authors describe precautions to protect the prosthesis from dislocation and acromial stress fractures, and propose a slow progressive approach to restoring motion and functional strength. The clinical guidelines published by these authors contrast with a very progressive criterion based rehabilitation plan that allows early use of the arm and very little immobilization. Neither of these two proposed rehabilitation plans are associated with clinical trials that track clinical or functional outcome measures or complication rate. A chapter devoted to rehabilitation following RSA in the book "Reverse Shoulder Arthroplasty" suggests that physician directed video-based rehabilitation may be just as effective as formal physical therapy. The author points out the need for randomized controlled trials to determine the need for physical therapy following a variety of shoulder surgeries. Clarifying the impact of formal clinic based PT intervention following RSA is important in determining the best plan of care for this population following surgery, while ensuring that there is not an increase in complications associated with the therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have RSA for cuff tear arthropathy, massive irreparable rotator cuff tear with pseudoparalysis, or primary osteoarthritis.

Exclusion Criteria:

* Subjects who have a non-reverse total shoulder arthroplasty, RSA for fracture, tendon transfers as part of RSA, and revision RSA
* Subjects who had RSA and require discharge to skilled nursing facility, in-patient rehabilitation placement, or use of home health therapy prior to progressing in recovery
* Subjects who cannot speak, read, or write the English language
* Subjects who have cognitive deficits limiting ability to follow directions
* Subjects who have inability to attend physical therapy (i.e. transportation or financial limitations)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2025-08-11 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain: Numerical Rating Scale | up to 2 years postoperatively
  Pain measured using 0-10 Numeric Pain Rating Scale (NRS) with 0 being a better score
Range of motion | up to two years postoperatively
  Clinician measure of function using active and passive forward elevation, external rotation with the arm at the side in adduction and at 90 degrees of abduction in the scapular plane, and active internal rotation measured by highest vertebral level reached with thumb
Patient-reported functional outcome- American Shoulder and Elbow Surgeons Score | up to two years postoperatively
  American Shoulder and Elbow Surgeons (ASES). Survey is scored 0 to 100 with 0 being the lowest possible score indicating a poor outcome and 100 being the highest possible score and indicating a good outcome.
Patient-reported functional outcome- Single Assessment Numeric Evaluation score | up to two years postoperatively
  Single Assessment Numeric Evaluation (SANE) score. Survey is scored 0 to 100 with 0 being the lowest possible score indicating a poor outcome and 100 being the highest possible score and indicating a good outcome.

SECONDARY OUTCOMES:
Complication rates | up to 2 years postoperatively
  acromial stress fractures and shoulder dislocations monitored by patient report through phone calls, patient visits, clinical exams, and standard of care imaging. All complications will be combined as a composite measure.
Cost of Care | up to 2 years after surgery
  reimbursement for therapy services, total number of therapy visits, estimated travel time per visit, and associated costs. These measures will be combined in a cost-effectiveness analysis with a decision tree model.
Quality adjusted life years: PROMIS-29 | up to 2 years postoperatively
  assessed using Patient-Reported Outcomes Measurement Information System-29. PROMIS Profile instruments are a collection of short forms containing a fixed number of items from seven PROMIS domains (Depression, Anxiety, Physical Function, Pain Interference, Fatigue, Sleep Disturbance, and Ability to Participate in Social Roles and Activities).The PROMIS-29 assesses each of the 7 domains with 4 questions. Each of the 7 domains has a raw score range from 4 to 20 with 4 being the lowest score, indicating a poor outcome and 20 being the highest score, indicating a good outcome.(PROMIS-29) surveys
Postoperative Pain Medication Use Duration | up to two years postoperatively
  duration of narcotic medication usage as documented in the Illinois Prescription Monitoring Program (Illinois PMP) or equivalent monitoring program for non-Rush centers
Postoperative Pain Medication Prescription Refills | up to two years postoperatively
  number of narcotic medication prescription refills as documented in the Illinois Prescription Monitoring Program (Illinois PMP) or equivalent monitoring program for non-Rush centers

CONTACTS AND LOCATIONS:
Overall Officials: Grant E Garrigues, MD, Principal Investigator — Rush University Medical Center
Locations (7):
- United States (7):
  - Western Orthopaedics, Denver, Colorado
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - Rush University Medical Center, Chicago, Illinois
  - Centers for Advanced Orthopaedics, Leonardtown, Maryland
  - New England Baptist Hospital, Dedham, Massachusetts
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Anderson Orthopedic Clinic, Arlington, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ecklund KJ, Lee TQ, Tibone J, Gupta R. Rotator cuff tear arthropathy. J Am Acad Orthop Surg. 2007 Jun;15(6):340-9. doi: 10.5435/00124635-200706000-00003. PMID 17548883
- [Background] Schairer WW, Nwachukwu BU, Lyman S, Craig EV, Gulotta LV. National utilization of reverse total shoulder arthroplasty in the United States. J Shoulder Elbow Surg. 2015 Jan;24(1):91-7. doi: 10.1016/j.jse.2014.08.026. Epub 2014 Oct 29. PMID 25440519
- [Background] Berliner JL, Regalado-Magdos A, Ma CB, Feeley BT. Biomechanics of reverse total shoulder arthroplasty. J Shoulder Elbow Surg. 2015 Jan;24(1):150-60. doi: 10.1016/j.jse.2014.08.003. Epub 2014 Oct 29. PMID 25441574
- [Background] Boileau P, Watkinson DJ, Hatzidakis AM, Balg F. Grammont reverse prosthesis: design, rationale, and biomechanics. J Shoulder Elbow Surg. 2005 Jan-Feb;14(1 Suppl S):147S-161S. doi: 10.1016/j.jse.2004.10.006. PMID 15726075
- [Background] Samitier G, Alentorn-Geli E, Torrens C, Wright TW. Reverse shoulder arthroplasty. Part 1: Systematic review of clinical and functional outcomes. Int J Shoulder Surg. 2015 Jan-Mar;9(1):24-31. doi: 10.4103/0973-6042.150226. PMID 25709242
- [Background] Farshad M, Gerber C. Reverse total shoulder arthroplasty-from the most to the least common complication. Int Orthop. 2010 Dec;34(8):1075-82. doi: 10.1007/s00264-010-1125-2. Epub 2010 Sep 25. PMID 20865260
- [Background] Alentorn-Geli E, Samitier G, Torrens C, Wright TW. Reverse shoulder arthroplasty. Part 2: Systematic review of reoperations, revisions, problems, and complications. Int J Shoulder Surg. 2015 Apr-Jun;9(2):60-7. doi: 10.4103/0973-6042.154771. PMID 25937717
- [Background] Boudreau S, Boudreau ED, Higgins LD, Wilcox RB 3rd. Rehabilitation following reverse total shoulder arthroplasty. J Orthop Sports Phys Ther. 2007 Dec;37(12):734-43. doi: 10.2519/jospt.2007.2562. Epub 2007 Aug 28. PMID 18560182
- [Derived] Kennedy JS, Reinke EK, Friedman LGM, Cook C, Forsythe B, Gillespie R, Hatzidakis A, Jawa A, Johnston P, Nagda S, Nicholson G, Sears B, Wiesel B, Garrigues GE; SHORT Trial Investigators; Hagen C, Hong I, Roach M, Jones N, Mahendraraj K, Michaelson E, Bader J, Mauter L, Mengers S, Renko N, Strony J, Hart P, Steele E, Naylor A, Gaudette J, Sprengel K. Protocol for a multicenter, randomised controlled trial of surgeon-directed home therapy vs. outpatient rehabilitation by physical therapists for reverse total shoulder arthroplasty: the SHORT trial. Arch Physiother. 2021 Dec 10;11(1):28. doi: 10.1186/s40945-021-00121-2. PMID 34886910